CLINICAL TRIAL: NCT03921099
Title: Evaluation of the Impact of Ascorbic Acid in the Prevention of Vancomycin Induced Nephrotoxicity
Brief Title: Impact of Ascorbic Acid in the Prevention of Vancomycin Induced Nephrotoxicty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Nouran Hesham Ali, clinical pharmacist at the critical care medicine unit- Cairo university hospitals, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 208
Record Dates: First submitted 2019-04-16; First posted 2019-04-19 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vancomycin only (No Intervention): Vancomycin 15-20mg/kg intravenous every 8-12 hours.
- Vancomycin +Ascorbic acid (Experimental): Vancomycin 15-20mg/kg intravenous every 8-12 hours. Ascorbic acid 1gm every 12 hours orally just before vancomycin by half an hour for seven days.
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — ascorbic acid is an antioxidant that is expected to prevent nephrotoxicty induced by Vancomycin.
  Other Names: Vitamin C
  Arms: Vancomycin +Ascorbic acid

SUMMARY:
A Randomized controlled trial aiming to investigate whether ascorbic acid has a role in preventing vancomycin induced nephrotoxicity or not in critically ill patients.

DETAILED DESCRIPTION:
Critically ill patients who have gram positive infection (MRSA) and need vancomycin will be assigned randomly into two groups. The first group will be given vancomycin intravenous only (15-20 mg/kg) every 8-12 hours , while the second group will take vancomycin intravenous (15-20 mg/kg) every 8-12 hours plus ascorbic acid 1 gram twice daily orally just before the vancomycin administration by half an hour. Patients will be monitored for one week where serum creatinine, BUN, urine output, trough level will be measured. Acute kidney injury will be determined according to RIFLE criteria.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are critically ill and with MRSA infection suspection.

Exclusion Criteria:

1. Pregnancy or breast feeding.
2. Known allergy to either vancomycin or ascorbic acid.
3. Base line serum creatinine ≥2mg/dl.
4. Patients receiving other nephrotoxic drug (e.g., aminoglycosides, amphotericin B, cisplatin or calcinurine inhibitors).
5. Anticepated administration of contrast medium within 7 days.
6. Patients suffering from some underlying diseases (e.g., cancer, HIV infection, systemic lupus erythematoses,or urinary tract stones).
7. Unlikelyhood of receiving the study medications for at least 72 hours

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of nephrotoxicty | one week
  Incidence of nephrotoxicty will be described according to RIFLE criteria

SECONDARY OUTCOMES:
28 days Mortality | one month

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa A Sabry, PhD, Study Director — Ain Shams University; Sara M Shaheen, PhD, Study Director — Ain Shams University
Locations (1):
- Cairo university hospitals, Cairo, Egypt

REFERENCES:
- [Derived] Hesham El-Sherazy N, Samir Bazan N, Mahmoud Shaheen S, A Sabri N. Impact of ascorbic acid in reducing the incidence of vancomycin associated nephrotoxicity in critically ill patients: A preliminary randomized controlled trial. F1000Res. 2021 Sep 16;10:929. doi: 10.12688/f1000research.55619.1. eCollection 2021. PMID 34621519